CLINICAL TRIAL: NCT01760746
Title: A Randomized, Multi-Centre, Double-Masked, Study to Compare Inflammatory Protein Changes in Aqueous Humour of Subjects Treated With Bevacizumab (Avastin) vs Ranibizumab (Lucentis) Pre-Vitrectomy for Proliferative Diabetic Retinopathy
Brief Title: Comparison of Changes of Inflammatory Proteins in Aqueous Humour of Subjects Treated With Avastin vs Lucentis
Acronym: Humour
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H11-02704
Record Dates: First submitted 2012-12-14; First posted 2013-01-04 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Proliferative Diabetic Retinopathy (PDR)
Keywords: Proliferative Diabetic Retinopathy; Vitrectomy; Inflammatory Cytokines
MeSH Terms: interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humour
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PDR, Avastin/Lucentis, randomization, humour, inflamation: Patients will be randomized to receive pre-treatment with either bevacizumab or ranibizumab . Sample of aqueous humour will be taken before injection and before surgery.Both the patient and the treating physician will be masked to the identity of the study drug.
  Interventions: Other: Injection of Avastin / Lucentis, sampling aqueous humour

INTERVENTIONS:
Other: Injection of Avastin / Lucentis, sampling aqueous humour — Study participants will be divided into two arms. Subjects will receive Avastin or Lucentis a few days before vitrectomy surgery. The assignment will be double-masked.The first sample of aqueous humor will be obtained immediately prior to the intravitreal injection.
  On the same of the intravitreal injection, a blood sample will be taken for hemoglobin A1C measurement. Approximately 1 week later when patients are having their scheduled vitrectomy surgery, an additional sample of aqueous humour will be obtained .
  Intraocular cytokines levels will be measured in aqueous humor samples using multiplex cytokine assays.
  Other Names: Humour; Inflamatory Cytokines; Avastin; Lucentis

SUMMARY:
PDR is a leading cause of irreversible vision loss in North America. This disease is caused by the growth of abnormal blood vessels in the retina. These abnormal blood vessels can bleed inside the eye, causing a vitreous hemorrhage (VH). Sometimes when patients have this bleeding, a surgery called vitrectomy is required to remove the blood from within the eye. In order to reduce complications during the surgery, most retina surgeons will inject Avastin into the eye a few days before the surgery.

Avastin (bevacizumab) is currently not approved by Health Canada to treat any ocular disease. Lucentis (ranibizumab) is approved by Health Canada as a treatment for age-related macular degeneration, diabetic macular edema, and retinal venous occlusive disease. While Avastin is not approved by Health Canada for the treatment of these diseases, the majority of retina specialists around the world are now using Avastin "off-label" to treat these diseases. That is because Avastin and Lucentis both tend to work equally well in these disease, but Avastin is significantly cheaper. While Avastin and Lucentis are generally regarded to be equal, there may be some differences between these two drugs that have not been discovered. The aim of this study is to look for these differences.

Previous research by the investigators in this study has shown that injecting Avastin into eyes causes increased inflammatory proteins to develop inside the eye. This increase in these proteins was related to complications that developed after the vitrectomy surgery. Lucentis may be associated with less of an increase in inflammatory proteins (and less complications). The aim of this study will be to compare Avastin and Lucentis with respect to how they affect inflammatory proteins in the eye, as well as the rate of complications during surgery.

Study participants will be divided into two arms ("groups") of 30 subjects. Subjects will receive Avastin or Lucentis a few days before vitrectomy surgery. The assignment will be random and the study is double-masked. Masking is done so that the investigators can clearly determine any differences between the 2 drugs.

DETAILED DESCRIPTION:
60 subjects will take part in this study at 2 sites in Canada: Vancouver (Eye Care Centre, Vancouver General Hospital, and Mount Saint Joseph Hospital) and Toronto (Sunnybrook Health Sciences Centre).

ELIGIBILITY:
Inclusion Criteria:

1. PDR and vitreous hemorrhage scheduled for vitrectomy surgery and bevacizumab pre-treatment.

Exclusion criteria:

1. Vitreous hemorrhage from other causes such as central retinal vein occlusion or ocular ischemic syndrome.
2. Pregnant or breastfeeding women.
3. Less than 19 years of age.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to assess changes in intraocular levels of cytokines following anti-VEGF treatment, the ideal time to measure these cytokines is at baseline and approximately 1 week later. In patients with PDR who are scheduled for vitrectomy, many vitreoretinal surgeons now inject bevacizumab approximately 1 week prior to the surgery in order to decrease the risk of intra-operative complications. These patients are thus an excellent study group for studying intraocular cytokine changes in response to anti-VEGF therapy, since that are already scheduled to have 2 intraocular procedures performed approximately 1 week apart, thereby minimizing the risk of obtaining aqueous humour.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in global levels of intraocular inflammatory cytokines in the aqueous humour of patients with Proliferative Diabetic Retinopathy. | Baseline and two weeks
  No single inflammatory cytokine or any summary measure of the cytokines has been shown to characterize the effect of anti-VEGF (Vascular Endothelial Growth Factor)treatment; therefore, we will employ a global test to compare the difference of all inflammatory cytokines between the two treatment groups. For each cytokine the endpoint will be defined as percentage change from baseline. We will employ O'Brien's rank-sum global test to simultaneously evaluate all the inflammatory cytokine endpoints. O'Brien's test is a nonparametric test procedure for testing whether multiple outcomes in one treatment group have consistently larger values than outcomes in the other treatment group.

SECONDARY OUTCOMES:
Secondary outcomes include the change in angiogenic cytokine levels. | Baseline and two weeks
  Study outcomes will be analyzed using multivariate models, and covariates will include age, gender, diabetes type, hemoglobin A1C (glycosilated hemoglobin)level, and the number of days between the time of anti-VEGF pretreatment and vitrectomy.
Secondary outcome measure considers intraoperative complications during vitrectomy. | Baseline and two weeks
  The following intra-operative data will be recorded: use of adjunctive intravitreal/periocular triamcinolone (Kenalog®,)presence of tractional retinal detachment, occurrence of intra-operative bleeding and iatrogenic tears, use of endodiathermy/endolaser, and mean surgical time.

CONTACTS AND LOCATIONS:
Overall Officials: Farzin Forooghian, MD FRCSC, Principal Investigator — Clinical Assistant Professor
Locations (1):
- UBC/VGH Eye Care Centre, Vancouver, British Columbia, Canada